CLINICAL TRIAL: NCT05808621
Title: Investigation of Peripheral Muscle Oxygenation at Rest and Movement in Hospitalized Patients in Severe Acute Exacerbation of Chronic Obstructive Pulmonary Disease and Comparison With Stable Period
Brief Title: Muscle Oxygenation in Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Gulhan Yilmaz Gokmen, Assistant Professor, Bandırma Onyedi Eylül University
Other Study IDs: 2023-19
Record Dates: First submitted 2023-03-13; First posted 2023-04-11 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Chronic Obstructive Pulmonary Disease Exacerbation; Muscle Oxygenation
Keywords: Chronic Obstructive Pulmonary Disease; Muscle Oxygenation; Chronic Obstructive Pulmonary Disease Exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of our study is to examine the Peripheral Muscle Oxygenations at rest and in motion on the 2nd day of hospitalized patients and before discharge in Severe Acute Exacerbation of Chronic Obstructive Pulmonary Disease and to compare the results in the hospital periods by repeating the tests in the stable periods of the patients 1 month after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Being a COPD patient hospitalized with Severe Acute Exacerbation
* be between 40-80 years old
* Having a Body Mass Index below 35

Exclusion Criteria:

* Patients who do not want to participate in the study
* Patients requiring intensive care follow-up during their hospitalization Arthritis, neurological disease, deep vein thrombosis, peripheral arterial disease, muscle weakness, broken etc. patients with the condition
* Extensive parenchyma such as malignancy, pulmonary embolism, vasculitis, collagen tissue diseases, interstitial fibrosis, severe pneumonia patients with damage
* Patients with severe dyspnea and hemodynamic instability who cannot perform the sit-up test

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD hospitalized with Severe Acute Exacerbation
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-06-23 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Muscle oxygenation | 4 weeks
  The muscle oxygen monitor is a lightweight (42 g) and small (dimensions: 61 × 44 × 21 mm) device that measures regional blood flow and oxygenation by placing it on the skin non-invasively with near infrared spectroscopy (NIRS). The device, which has data collection and telemetric features, also allows O 2 measurement in non-laboratory environments and field-based research.

SECONDARY OUTCOMES:
1 minute sit and stand test | 4 weeks
  The test aims to assess your exercise capacity and leg muscle strength. The movement required is to get up from this chair with the legs straight and sit back continuing the repetitions as fast as possible within one minute.
  The 1-minute STS test was performed with a chair of standard height of 46 cm without armrests. The patient was ensured to be seated upright on the chair positioned against a wall. The patient sat with the knees and hips flexed to 90°, feet placed flat on the floor hip-width apart, and the hands placed on the hips. Every get up from one's chair was validated to check if a complete sit-to-stand-to-sit sequence was achieved.
Modified Medical Research Council Dyspnea Scale: | 4 weeks
  Medical Research Council (MRC) Dyspnea Scale will be used to assess the severity of dyspnea. The severity of dyspnea during activities of daily living is graded from 0 to 4 on the Medical Research Council (MRC) Dyspnea Scale.
COPD Assessment Test (CAT) | 4 weeks
  The COPD Assessment Test (CAT) is a new scoring system for COPD patients, which provides a simple method for assessing the impact of COPD on the patient's health. Range of CAT scores from 0-40.
Charlson Comorbidity Index | 4 weeks
  The Charlson Comorbidity Index was first developed in 1987 by Mary Charlson and colleagues as a weighted index to predict risk of death within 1 year of hospitalization for patients with specific comorbid conditions. Nineteen conditions were included in the index. The total score in the CCI is derived by summing the assigned weights of all comorbid conditions presented by the client. Higher scores indicate a more severe condition and consequently, a worse prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma Onyedi Eylül University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No